CLINICAL TRIAL: NCT06154746
Title: Analysis of Risk Factors in the Development of Diabetic Retinopathy in Assuit University Hospital
Brief Title: Analysis of Risk Factors of Diabetic Retinopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dalia Mohamed Mahmoud Asem, resident doctor, Assiut University
Other Study IDs: risk factors of DR
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: slit lamb & OCT — 1. The Slit lamb is a biomicroscope. It emits a beam of light that can be varied in height and width. It allows visualization of the anterior segment of the eye. With auxiliary lenses, the examiner can also view the posterior segment. These lenses are simple, affordable, and portable. Although high-end devices like fundus cameras and optical coherence tomography have revolutionized how practitioners detect eye diseases, they can never replace these handheld lenses.
  2. OCT is a noninvasive method that yields a cross-section image of the retina by exposing the eye to near-infrared light. Specifically, an emitted light beam is scattered and reflected back by the retinal surface as well as its different layers.

SUMMARY:
The aim of the study is to analyse the risk factors involved in the development of diabetic retinopathy.

DETAILED DESCRIPTION:
Introduction Worldwide, diabetic retinopathy (DR) is the leading cause of blindness among working age adults [1]

Diabetes mellitus (diabetes) is a group of conditions in which elevation and dysregulation of blood glucose levels result from either decreased production of insulin or systemic resistance to insulin's effects.

Economic costs of diabetes in the. U.S. in 2012. Diabetes Care. 2013;36(4):1033-46.

Insulin resistance, which often precedes type 2 diabetes, is a component of the metabolic syndrome. Those with diabetes are more likely to have other components of the metabolic syndrome including abdominal obesity, dyslipidemia, hypertension, prothrombotic state, and a proinflammatory state [2] Third Report of the National Cholesterol Education Program. (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002;106(25):3143-421

Another key point for the development of vascular lesions is the capillary basement membrane thickening as a result of hyperglycemia, increased synthesis of basement membrane components and other factors. This thickening of the basement membrane is related to excess vascular permeability that leads to leaky vessels, compromised tight-junctions and increased vesicular transport [3]

Although major risk factors-hyperglycemia and hypertension-are extensively studied and show a strong association with DR

Some studies indicate that prolonged DM duration is indeed a well-established risk factor for DR [4-5]. Regarding microalbuminuria, studies report its association as a marker of microvascular dysfunction and DR [6-7], however further studies are needed to confirm this relationship [6]. Other risk factors such as body mass index (BMI) show controversies in relation to its association with this disease [8]. The aim of this study was to investigate risk factors for DR.

Diabetic retinopathy is the leading cause of blindness in adults living in developed countries.9 Almost all patients with type 1 diabetes mellitus (DM) and more than 60% of patients with type 2 DM will develop some degree of retinopathy after a 20-year history of diabetes.10 It has also been well established that DM increases the risk of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

All patients with confirmed DR , best-corrected visual acuity BCVA (using a Snellen chart) in each eye to allow the performance of the protocol, and intraocular pressure less than 21 mmHg.

• . proliferative diabetic retinopathy with or without high-risk characteristics (HRCs) (any three of the following):

* presence of neovessels
* location of the neovessels (at the optic nerve)
* size of the neovessels: if at the optic nerve [neovascularisation of the disc (NVD)] ≥ ¼-⅓ disc area if elsewhere in the retina [neovascularisation of the retina elsewhere (outside the disc) (NVE) ≥ ½ of the disc area (if both NVD and NVE present, classified based on neovessels at the disc)
* presence of pre-retinal haemorrhage or vitreous haemorrhage. About half of patients with severe or very severe NPDR will progress to PDR within a year.

Symptoms include sudden de crease of V/A , appearance of flashes and floaters, visual field defects.

Exclusion Criteria:

* The exclusion criteria were: DM other than T2DM (such as gestational diabetes); known severe mental illness; a separate advanced or terminal condition; and severe advanced diabetic complications defined as being registered blind, requiring dialysis, or having had an above-the-knee amputation

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population-based, cross-sectional survey using the standardised Rapid Assessment of Avoidable Blindness with the addition of the Diabetic Retinopathy module methodology.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
aeffect of risk factors in progression of diabetic retinopathy. | baseline
  analysis of risk factors affecting progression of diabetic retinopathy and test if they can be modified or not.